CLINICAL TRIAL: NCT00732238
Title: Multifaceted Treatment of Catheter-related Urinary Tract Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B4747-P; H-18309 (Other Grant/Funding Number: Baylor College of Medicine)
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Spinal Cord Injury; Neurogenic Bladder; Urinary Tract Infection
Keywords: Spinal Cord Injury; Urinary Tract Infection; Catheter Dependent
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Tract Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Removal of Bladder Catheter. Urine Culture Post Catheter Removal. Shorter Duration of Antibiotic Therapy.
  Interventions: Other: Shortened course of antibiotic therapy
- Arm 2 (Active Comparator): Urinary Catheter Is Not Exchanged. Antibiotic Therapy Is Based On Culture Obtained From Existing Catheter. Longer Duration of Antibiotic Therapy.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Other: Shortened course of antibiotic therapy — By obtaining a urine culture from a newly inserted catheter we hope to find the true urinary pathogen. In so doing we feel a shorter but pathogen specific course of antibiotic therapy will more successfully prevent urinary tract infection relapse.
  Arms: Arm 1
Other: Standard Therapy — Patients entered into this arm of the study will receive the standard duration of antibiotic therapy, which will be determined by urine culture results obtained from existing urinary catheter.
  Arms: Arm 2

SUMMARY:
The specific objective of this clinical trial is to demonstrate that a multifaceted approach for treatment for catheter-related urinary tract infection (UTI) in patients with spinal cord injury is effective and feasible. We plan to test the following hypothesis: a multifaceted treatment approach that consists of immediate removal of the indwelling bladder catheter, selecting antibiotics based on the finding from a urine culture that is obtained through the newly inserted catheter, and a 5-day course of systemic antibiotics will effectively treat catheter-related infection that is limited to the lower urinary tract of patients with spinal cord injury.

DETAILED DESCRIPTION:
UTI is the most common infection in patients with spinal cord injury who require a catheter to drain urine from their bladder. These infections can cause serious medical complications, such as bloodstream infection, decreased kidney function, prolonged hospitalization, and add great cost. Unfortunately, the treatment of catheter-related urinary tract infection has not been standardized in this population in terms of:

* the need to replace the indwelling catheter;
* the necessity to provide antibiotic coverage against all organisms grown from urine cultures; and
* the duration of antibiotic treatment.

The prevalent, though not scientifically well supported approach for treating catheter-related lower UTI in patients with spinal cord injury comprises the following:

* Retaining the original bladder catheter in place upon diagnosis of infection because of the theoretical concern that removal of the infected catheter may potentially cause the infecting organism to move from the bladder to the bloodstream (bacteremia). This theoretical complication, however, is very unlikely and even if it does occur, the bacteria would only remain in the bloodstream for a very short period of time and would not have a significant impact on the patient. In contrast, we propose that immediate removal of the original indwelling bladder catheter with its film of protected bacteria can enhance resolution of UTI.
* Providing antibiotic coverage against all organisms which grow from a urine culture that is obtained from the original indwelling bladder catheter. Although this source of urine culture is a sensitive method for identifying the organisms that are present in the urine, it suffers from poor specificity because it may yield the growth of some organisms that could have colonized the catheter (and, therefore, grown in a culture of urine obtained through that original catheter) but did not contribute to UTI. This issue is particularly problematic in patients with spinal cord injury because urine cultures in almost half of the cases of UTI in this population yield multiple bacteria. Therefore, we propose that collection of a urine culture while inserting the new bladder catheter would yield growth of only organisms that truly contribute to UTI and, therefore, obviate the need to administer unnecessary antibiotics to cover additional organisms that would grow only from urine cultures obtained through the original catheter.
* Treatment with systemic antibiotics for 10 days. There exists, however, no prospective randomized clinical trials indicating that this duration of antibiotic therapy is optimal in patients with spinal cord injury. Since catheter-free, able-bodied patients with lower UTI are successfully treated with courses of antibiotics as short as 1-3 days, we propose that by removing the focus of infection (i.e. the original catheter) a 5-day course of systemic antibiotics would be sufficient for treating catheter-related lower UTI in patients with spinal cord injury.

The results of this research are expected to provide the following major benefits to veterans with spinal cord injury:

* the multifaceted approach will provide highly effective treatment of UTI;
* the lower number of antibiotics that are administered to cover the organisms grown from urine cultures obtained at the time of inserting the replacement bladder catheter will result in lower cost of treatment and a reduced risk for developing antibiotic resistance;
* the shorter duration of antibiotic course will decrease the overall cost of treatment, reduce hospital stay, and shorten rehabilitation down time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with SCI who are hospitalized at the Michael E. Debakey VA Medical Center and suffer from lower UTI associate with an indwelling transurethral or suprapubic bladder catheter will be enrolled in the study

Exclusion Criteria:

* Exclusion criteria will include septicemia, chronic antimicrobial therapy and inability, or unwillingness to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih O Darouiche, MD, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- New Catheter Arm: Removal of Bladder Catheter. Urine Culture Post Catheter Removal. Shorter Duration of Antibiotic Therapy.
  Shortened course of antibiotic therapy: By obtaining a urine culture from a newly inserted catheter we hope to find the true urinary pathogen. In so doing we feel a shorter but pathogen specific course of antibiotic therapy will more successfully prevent urinary tract infection relapse.
- Existing Catheter Arm: Urinary Catheter Is Not Exchanged. Antibiotic Therapy Is Based On Culture Obtained From Existing Catheter. Longer Duration of Antibiotic Therapy.
  Standard Therapy: Patients entered into this arm of the study will receive the standard duration of antibiotic therapy, which will be determined by urine culture results obtained from existing urinary catheter.
Period: Overall Study
Arm/Group | New Catheter Arm | Existing Catheter Arm
Started | 33 | 28
Completed | 28 | 27
Not Completed | 5 | 1
Not completed — Bacteremia | 4 | 1
Not completed — Asymptomatic bacteriuria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Catheter Arm | Existing Catheter Arm | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (13) | 58.3 (14.8) | 59.9 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 25 | 27 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 16 | 14 | 30
  Black | 11 | 13 | 24
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Outcome of the Study is Response to Treatment Which Will be Assessed at the End of Therapy. Successful Response to Treatment is Defined as Resolution of Clinical Manifestations of Infection Plus Lack of Growth of the Original Infect
Time Frame: Patients will be evaluated for signs of continued infection at mid therapy and at the end of antibiotic therapy (day 5 for new catheter arm and day 10 for existing catheter arm)
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 28 | 27
participants | 28 | 27

2. Secondary Outcome: The Secondary Efficacy Outcome is Recurrence of UTI up to 180 Days After the End of Therapy
Description: Relapse of UTI is defined as a recurrence of clinical manifestations of infection plus growth of the original infecting pathogen(s) in urine culture in association with significant pyuria (>10 WBC/phf)
Time Frame: Up to 180 days of end of therapy
Measure: Number; unit: participants
Arm/Group | New Catheter Arm | Existing Catheter Arm
Number analyzed (Participants) | 28 | 27
participants | 9 | 3

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 2/28 | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=28) | Arm 2 (N=27)
C diff colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes